CLINICAL TRIAL: NCT04772755
Title: Preventing Post-Vaccination Presyncope and Syncope in Adolescents Using Simple, Clinic-based Interventions
Brief Title: Presyncope (Syncope) Prevention Study
Acronym: PS^2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00107635
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Syncope, Vasovagal
Keywords: Adolescent; Child; Buzzy®; Electronic Game; Syncope; Pain Mitigation; Anxiety; Presyncope; Vaccination; Syncope Prevention
MeSH Terms: conditions — Syncope, Vasovagal; Syncope; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants received usual care that followed administration of a vaccine and a 20 minute post vaccination observation period.
- Buzzy ® and Electronic Game (Experimental): Buzzy® was applied to the arm receiving vaccination for 30-60 seconds prior to vaccination and removed following vaccination. For the electronic game, participants were instructed to select a game from a prepopulated list of games on a tablet provided by the study team and then played that game for a specified amount of time before, during and after the vaccination administration.
  Interventions: Device: Buzzy® and Electronic Game

INTERVENTIONS:
Device: Buzzy® and Electronic Game — Buzzy® was applied according to manufacturers directions and an electronic game was played. The participant was observed for 20 minutes post vaccination.
  Arms: Buzzy ® and Electronic Game

SUMMARY:
This study was a prospective, randomized clinical trial that was conducted in adolescents (10 through 14 years of age) receiving at least one recommended intramuscularly administered vaccine to evaluate the efficacy and acceptability of using two different, simultaneously administered interventions that might prevent post-vaccination presyncope, and by extension syncope. The two interventions evaluated together were Buzzy®, which is a medical device designed to reduce vaccination pain, and an electronic game. The investigators evaluated both interventions when administered simultaneously (Buzzy® and electronic game). The investigators enrolled approximately 340 subjects into this study. Eligible adolescents were randomized (1:1) to either the intervention or control group: 1) intervention (Buzzy® and electronic game); or 2) control (usual care) to assess for acceptability and efficacy. Detailed data were collected and described from study participants including demographics, medical history, baseline generalized and state anxiety, and needle phobia. Participants were observed for 20 minutes following receipt of vaccines and reassessed for post-vaccination state anxiety, immediate and subsequent post-vaccination pain (within 1 minute and at 10 minutes), and the occurrence of witnessed syncope or presyncope, and presyncopal symptoms as rated by the modified Blood Donation Reactions Inventory (BDRI). Participants were asked to assess their acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 10 years through 14 years of age
2. The subject must be receiving at least one vaccine delivered intramuscularly
3. The parent/guardian must be willing and capable of providing written informed consent for the adolescent and the adolescent must be willing and capable of providing assent.
4. The subject must be willing to stay for the completion of all study-related activities.
5. Parent/guardian and adolescent must speak and read English by self-report
6. Parent/guardian must be willing to let their child select an electronic game to play during the study

Exclusion Criteria:

1. Receipt of investigational or experimental vaccine or medication within the previous two weeks
2. Receipt of routine injectable medication
3. Permanent indwelling venous catheter
4. Blood drawn within the past hour or scheduled for a blood draw during the post-vaccination observation period
5. Injection of medication during the past hour or scheduled for injection of medication during the observation period.
6. Cold intolerance or cold urticaria
7. Raynaud's phenomenon
8. Sickle cell disease
9. Significant visual impairment or blindness
10. Significant auditory impairment or deafness
11. Febrile (>38.0°C) or acutely ill individuals
12. Upper arm or shoulder pain or injury
13. Video game-induced seizures
14. Adolescent or parent/Guardian is an immediate relative of study staff or an employee who is supervised by study staff.
15. Any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 338 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanual B Walter, MD, MPH, Principal Investigator — Duke University; Theresa Harrington, MD, Principal Investigator — Centers for Disease Control and Prevention; Karen R Broder, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Participants received usual care that follows administration of a vaccine and a 20 minute post vaccination observation period.
- Buzzy ® and Electronic Game: Buzzy® was applied to the arm receiving vaccination for 30-60 seconds prior to vaccination and removed following vaccination. For the electronic game, participants were instructed to select a game from a prepopulated list of games on a tablet provided by the study team and then play that game for a specified amount of time before, during and after the vaccination administration.
  Buzzy® and Electronic Game: Buzzy® were applied according to manufacturers directions and an electronic game was played. The participant was observed for 20 minutes post vaccination.
Period: Overall Study
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Started | 170 | 168
Completed | 167 | 165
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Randomized and subsequently determined to be ineligible | 2 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) analysis population is defined as those subjects who are enrolled, randomized into the study, and received an intramuscular vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Buzzy ® and Electronic Game | Total
Number analyzed (Participants) | 167 | 165 | 332
Age, Continuous [Mean (Full Range); unit: years] | 11.9 [10 to 14] | 11.8 [10 to 14] | 11.85 [10 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 87 | 173
  Male | 81 | 78 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 15 | 26
  Not Hispanic or Latino | 156 | 150 | 306
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 10 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 52 | 112
  White | 92 | 87 | 179
  More than one race | 3 | 17 | 20
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 167 | 165 | 332

OUTCOME MEASURES:

1. Primary Outcome: Number of Adolescents With Presyncope or Syncope After Vaccination in the Intervention and Usual Care Groups.
Description: Subjects were asked to complete a presyncope symptoms assessment (Modified BDRI: Blood Donations Reactions Inventory) at 20 minutes post vaccination. The number of adolescents with presyncope or syncope as determined by the modified BRDR or witnessed presyncope or syncope.
Time Frame: Day 1, 20 minutes post vaccination
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
Participants | 80 | 59
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.0249, Chi-squared

2. Secondary Outcome: Categorical Change (Increase, Decrease, no Change) in Pre- and Post- Vaccination State Anxiety.
Description: Subjects completed the Youth Momentary Anxiety Checklist pre vaccination and 20 minutes post vaccination. Subjects completed a Likert scale anxiety metric [The Youth Momentary Anxiety Checklist (YMAC)], with 12 emotions ranging from 1-4 (1 is best/no anxiety and 4 is worse/highest anxiety) and 1 figure ranging from 1-5 (lowest to highest anxiety) and these 13 scores are added together for analysis. The best/lowest score is a 13 and the highest score is a 53, with the pre-vaccination total score minus the post-vaccination total score as the outcome of interest.
Time Frame: Day1: Pre-vaccination (baseline), Post-vaccination (20 minutes)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 163 | 164
Participants
  Increase | 28 | 28
  Decrease | 121 | 123
  No Change | 14 | 13
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.8918, Mantel Haenszel

3. Secondary Outcome: Numeric Change (Mean and Range) in Pre- Minus Post- Vaccination State Anxiety.
Description: Subjects were asked to complete the Youth Momentary Anxiety Checklist pre vaccination and 20 minutes post vaccination. Subjects completed a Likert scale anxiety metric [The Youth Momentary Anxiety Checklist (YMAC)], with 12 emotions ranging from 1-4 (1 is best/no anxiety and 4 is worse/highest anxiety) and 1 figure ranging from 1-5 (lowest to highest anxiety) and these 13 scores are added together for analysis. The best/lowest score is a 13 and the highest score is a 53, with the pre-vaccination total score minus the post-vaccination total score as the outcome of interest.
Time Frame: Day1: Pre-vaccination (baseline), Post-vaccination (20 minutes)
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
scores on a scale | 5.69 [-13 to 37] | 5.23 [-11 to 37]
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.6587, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mean Injection-site Pain Scores on the Wong-Baker Faces Pain Scale© at ≤ 1 Minute Following Vaccination.
Description: Subjects were asked to complete a pain assessment (The Wong-Baker Faces Pain Scale©) ≤ 1 minute after vaccination. The Wong-Baker Faces Pain Scale is a Likert scale with 6 levels (0,2,4,6,8,10) where 0 is no pain and 10 is the most pain.
Time Frame: Day 1, ≤ 1 minute after vaccination
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
scores on a scale | 3.26 [0 to 10] | 2.51 [0 to 10]
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.0059, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Adolescents Reporting an Injection Site Pain Score ≥ 2, on the Wong-Baker Faces Pain Scale©, ≤ 1 Minute Following Vaccination.
Description: as for outcome 4
Time Frame: Day 1, ≤ 1 minute following vaccination
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
Participants | 136 | 124
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.1647, Chi-squared

6. Secondary Outcome: Number of Adolescents Reporting an Injection Site Pain Score ≥ 4, on the Wong-Baker Faces Pain Scale©, ≤ 1 Minute Following Vaccination.
Description: as for outcome 4
Time Frame: Day 1, ≤ 1 minute following vaccination
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
Participants | 77 | 53
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.0090, Chi-squared

7. Secondary Outcome: Mean Injection-site Pain Scores on the Wong-Baker Faces Pain Scale© at (Approximately) 10 Minutes Following Vaccination.
Description: Subjects were asked to complete a pain assessment (The Wong-Baker Faces Pain Scale©) 10 minutes after vaccination. The Wong-Baker Faces Pain Scale is a Likert scale with 6 levels (0,2,4,6,8,10) where 0 is no pain and 10 is the most pain.
Time Frame: Day 1, (approximately) 10 minutes following vaccination
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
scores on a scale | 1.54 [0 to 10] | 1.09 [0 to 10]
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.0273, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Adolescents Reporting an Injection Site Pain Score ≥ 2, on the Wong-Baker Faces Pain Scale©, at (Approximately) 10 Minutes Following Vaccination.
Description: as for outcome 7
Time Frame: Day 1, (approximately) 10 minutes following vaccination
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
Participants | 84 | 65
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.0458, Chi-squared

9. Secondary Outcome: Number of Adolescents Reporting an Injection Site Pain Score ≥ 4, on the Wong-Baker Faces Pain Scale©, at (Approximately) 10 Minutes Following Vaccination.
Description: as for outcome 7
Time Frame: Day 1, (approximately) 10 minutes following vaccination
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Buzzy ® and Electronic Game
Number analyzed (Participants) | 167 | 165
Participants | 30 | 19
Statistical Analysis 1: Comparison: Usual Care vs Buzzy ® and Electronic Game; Test type: Superiority; p = 0.0976, Chi-squared

10. Secondary Outcome: Number of Adolescents Reporting Perceptions About Their Vaccination Experience Via an Acceptability Survey - Like or Dislike
Description: The Buzzy and electronic game acceptability survey consists of 11 items with varying responses.
Time Frame: Day 1, approximately 20 minutes post vaccination
Population: Does not apply to the Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy ® and Electronic Game
Number analyzed (Participants) | 165
Participants
  How much do you like having Buzzy on your arm(s) during the shot(s)?: Disliked very much | 4
  How much do you like having Buzzy on your arm(s) during the shot(s)?: Disliked a little | 16
  How much do you like having Buzzy on your arm(s) during the shot(s)?: Neither liked nor disliked | 28
  How much do you like having Buzzy on your arm(s) during the shot(s)?: Liked a little | 35
  How much do you like having Buzzy on your arm(s) during the shot(s)?: Liked very much | 76
  How much do you like having Buzzy on your arm(s) during the shot(s)?: Not sure | 6
  How much do you like playing a game during the shot(s)?: Disliked very much | 1
  How much do you like playing a game during the shot(s)?: Disliked a little | 0
  How much do you like playing a game during the shot(s)?: Neither liked nor disliked | 19
  How much do you like playing a game during the shot(s)?: Liked a little | 22
  How much do you like playing a game during the shot(s)?: Liked very much | 122
  How much do you like playing a game during the shot(s)?: Not sure | 1

11. Secondary Outcome: Number of Adolescents Reporting Perceptions About Their Vaccination Experience Via an Acceptability Survey - Difficult or Easy
Description: The Buzzy and electronic game acceptability survey consists of 11 items with varying responses.
Time Frame: Day 1, approximately 20 minutes post vaccination
Population: Does not apply to the Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy ® and Electronic Game
Number analyzed (Participants) | 165
Participants
  How difficult or easy was holding or having Buzzy held on your arm(s) during the shot(s)?: Very difficult | 1
  How difficult or easy was holding or having Buzzy held on your arm(s) during the shot(s)?: Somewhat difficult | 8
  How difficult or easy was holding or having Buzzy held on your arm(s) during the shot(s)?: Neither difficult nor easy | 15
  How difficult or easy was holding or having Buzzy held on your arm(s) during the shot(s)?: Somewhat easy | 23
  How difficult or easy was holding or having Buzzy held on your arm(s) during the shot(s)?: Very easy | 111
  How difficult or easy was holding or having Buzzy held on your arm(s) during the shot(s)?: Not sure | 7
  How difficult or easy was it to select and play the game?: Very difficult | 2
  How difficult or easy was it to select and play the game?: Somewhat difficult | 3
  How difficult or easy was it to select and play the game?: Neither difficult nor easy | 7
  How difficult or easy was it to select and play the game?: Somewhat easy | 21
  How difficult or easy was it to select and play the game?: Very easy | 129
  How difficult or easy was it to select and play the game?: Not sure | 3

12. Secondary Outcome: Number of Adolescents Reporting Perceptions About Their Vaccination Experience Via an Acceptability Survey - Comfortable or Uncomfortable
Description: The Buzzy and electronic game acceptability survey consists of 11 items with varying responses.
Time Frame: Day 1, approximately 20 minutes post vaccination
Population: Does not apply to the Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy ® and Electronic Game
Number analyzed (Participants) | 165
Participants
  How comfortable or uncomfortable was Buzzy on your arm(s) during the shot(s)?: Very uncomfortable | 11
  How comfortable or uncomfortable was Buzzy on your arm(s) during the shot(s)?: Somewhat uncomfortable | 34
  How comfortable or uncomfortable was Buzzy on your arm(s) during the shot(s)?: Neither comfortable nor uncomfortable | 16
  How comfortable or uncomfortable was Buzzy on your arm(s) during the shot(s)?: Somewhat comfortable | 47
  How comfortable or uncomfortable was Buzzy on your arm(s) during the shot(s)?: Very comfortable | 53
  How comfortable or uncomfortable was Buzzy on your arm(s) during the shot(s)?: Not sure | 4
  How comfortable or uncomfortable were you playing a game when receiving shots?: Very uncomfortable | 4
  How comfortable or uncomfortable were you playing a game when receiving shots?: Somewhat uncomfortable | 5
  How comfortable or uncomfortable were you playing a game when receiving shots?: Neither comfortable nor uncomfortable | 12
  How comfortable or uncomfortable were you playing a game when receiving shots?: Somewhat comfortable | 37
  How comfortable or uncomfortable were you playing a game when receiving shots?: Very comfortable | 100
  How comfortable or uncomfortable were you playing a game when receiving shots?: Not sure | 7

13. Secondary Outcome: Number of Adolescents Reporting Perceptions About Their Vaccination Experience Via an Acceptability Survey - Yes or no
Description: The Buzzy and electronic game acceptability survey consists of 11 items with varying responses.
Time Frame: Day 1, approximately 20 minutes post vaccination
Population: Does not apply to the Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy ® and Electronic Game
Number analyzed (Participants) | 165
Participants
  Did the cold temperature of Buzzy bother you?: No | 113
  Did the cold temperature of Buzzy bother you?: Yes | 35
  Did the cold temperature of Buzzy bother you?: Not sure | 17
  Did the vibration of Buzzy bother you?: No | 147
  Did the vibration of Buzzy bother you?: Yes | 10
  Did the vibration of Buzzy bother you?: Not sure | 8
  If you had the choice, would you like to use Buzzy again when receiving shot(s)?: No | 19
  If you had the choice, would you like to use Buzzy again when receiving shot(s)?: Yes | 131
  If you had the choice, would you like to use Buzzy again when receiving shot(s)?: Not sure | 15
  If you had the choice, would you like to play a game again when receiving shot(s)?: No | 18
  If you had the choice, would you like to play a game again when receiving shot(s)?: Yes | 134
  If you had the choice, would you like to play a game again when receiving shot(s)?: Not sure | 13

ADVERSE EVENTS:
Time Frame: During the 20-minute post-vaccination monitoring period
Description: Only Serious Adverse Events were collected during the 20-minute post-vaccination monitoring period; Other (Not Including Serious) Adverse Events were not collected.
Arm/Group | Usual Care | Buzzy ® and Electronic Game
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/165
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/165
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT04772755/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT04772755/SAP_002.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT04772755/ICF_000.pdf